CLINICAL TRIAL: NCT00055523
Title: A Phase II Study of the Human Anti-TNF Antibody Adalimumab for the Induction of Clinical Remission in Subjects With Crohn's Disease
Brief Title: A Study of the Human Anti-TNF Antibody Adalimumab for the Induction of Clinical Remission in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M02-403
Record Dates: First submitted 2003-03-04; First posted 2003-03-06 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab (D2E7)

SUMMARY:
Purpose of the study is to test whether adalimumab can induce clinical remission in subjects with active Crohn's disease when compared to placebo (an inactive substance)

ELIGIBILITY:
Inclusion:

* Diagnosis of Crohn's disease
* CDAI score at baseline of between 220 and 450
* Normal laboratory parameters
* Willing and able to give informed consent

Exclusion:

* Diagnosis of ulcerative colitis
* Women cannot be pregnant or breastfeeding
* No previous use of infliximab or other anti-TNF antagonists
* No previous history of tuberculosis or listeria infection
* No previous history of cancer other than successfully treated skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-04

PRIMARY OUTCOMES:
comparison of the induction of clinical remission
(achievement of a CDAI <150) of adalimumab 40 mg and 80 mg vs. placebo at Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Hanauer, MD, Principal Investigator — University of Chicago Department of Medicine
Locations (43):
- United States (43):
  - Gastroenterology Associates of the East Bay, Berkeley, California
  - Long Beach Gastroenterology Assoc., Long Beach, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Gastroenterology Assoc. of Fairfield Co., Bridgeport, Connecticut
  - Cleveland Clinic Florida, Weston, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Assoc., Atlanta, Georgia
  - Southeastern Digestive & Liver Disease, Savannah, Georgia
  - Northwest Gastroenterologists, S.C., Arlington Heights, Illinois
  - University of Chicago, Chicago, Illinois
  - Drug Research Services, Inc., Metairie, Louisiana
  - LSU School of Medicine, New Orleans, Louisiana
  - Digestive Disorders Associates, Annapolis, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Mayo Clinic and Mayo Foundation, Rochester, Minnesota
  - Gastroenterology and Hepatology, Kansas City, Missouri
  - Glenn Gordon, MD, Mexico, Missouri
  - Deaconess Billings Clinic Research Division, Billings, Montana
  - Gastroenterology Specialties, P.C., Lincoln, Nebraska
  - Long Island Clinical Research Associates, Great Neck, New York
  - NY Center for Clinical Research, Lake Success, New York
  - New York Presbyterian Hospital, New York, New York
  - Daniel Present, New York, New York
  - Rochester Institute for Digestive Diseases, Rochester, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Carolina Research Associates, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Oklahoma Foundation for Digestive Disease, Oklahoma City, Oklahoma
  - Research Solutions, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Peter Molloy, MD, Pittsburgh, Pennsylvania
  - Diseases of the Digestive System, Chattanooga, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Northwest Gastroenterology, Bellevue, Washington
  - Inland Empire Gastroenterology, Spokane, Washington
  - Tacoma Digestive Disease Center, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Steenholdt C, Al-khalaf M, Brynskov J, Bendtzen K, Thomsen OO, Ainsworth MA. Clinical implications of variations in anti-infliximab antibody levels in patients with inflammatory bowel disease. Inflamm Bowel Dis. 2012 Dec;18(12):2209-17. doi: 10.1002/ibd.22910. Epub 2012 Feb 16. PMID 22344964